CLINICAL TRIAL: NCT00791544
Title: Dose-finding, Safety, Pharmacokinetic and Pharmacodynamic Study of AVE1642, an Anti-Insulin-like Growth Factor-1 Receptor (IGF-1R/CD221) Monoclonal Antibody, Administered as Single Agent and in Combination With Other Anti Cancer Therapies (Sorafenib or Erlotinib) in Patients With Advanced Liver Carcinoma
Brief Title: Dose Finding Study of AVE1642 in Patients With Advanced or Metastatic Liver Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue the AVE1642 development program, not due to any safety or efficacy concerns
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED10630; EudraCT 2008-000809-10
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Liver Carcinoma
Keywords: monoclonal antibody, anti IGF1R
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — AVE1642; Sorafenib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Dose Level -1 (Experimental): 0.5 mg/kg AVE1642 single agent at cycle 1 with sorafenib at cycle 2
  Interventions: Drug: AVE1642; Drug: sorafenib
- Dose Level 1 (Experimental): 1 mg/kg AVE1642 single agent at cycle 1 with sorafenib at cycle 2
  Interventions: Drug: AVE1642; Drug: sorafenib
- Dose Level 2 (Experimental): 3 mg/kg AVE1642 single agent at cycle 1 with sorafenib at cycle 2
  Interventions: Drug: AVE1642; Drug: sorafenib
- Dose Level 3 (Experimental): 6 mg/kg AVE1642 single agent at cycle 1 with sorafenib at cycle 2
  Interventions: Drug: AVE1642; Drug: sorafenib
- Dose Level 4 (Experimental): 12 mg/kg AVE1642 single agent at cycle 1 with sorafenib at cycle 2
  Interventions: Drug: AVE1642; Drug: sorafenib
- Dose Level 5 (Experimental): 18 mg/kg AVE1642 single agent at cycle 1 with sorafenib at cycle 2
  Interventions: Drug: AVE1642; Drug: sorafenib
- Combination cohort 1 (Experimental): AVE1642 selected dose in combination with sorafenib
  Interventions: Drug: AVE1642; Drug: sorafenib
- Combination cohort 2 (Experimental): AVE1642 selected dose in combination with erlotinib
  Interventions: Drug: AVE1642; Drug: erlotinib

INTERVENTIONS:
Drug: AVE1642 — intravenous infusion
Drug: sorafenib — oral intake
  Other Names: Nevaxar
  Arms: Combination cohort 1; Dose Level -1; Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4; Dose Level 5
Drug: erlotinib — oral intake
  Other Names: Tarceva
  Arms: Combination cohort 2

SUMMARY:
The primary objective of the study is to select the dose of AVE1642 to be administered in patients with liver carcinoma not eligible for local treatment.

The secondary objectives of the study are:

* To evaluate the safety profile of AVE1642 as single agent and the safety profile of combinations with other anti-cancer therapies of interest in liver carcinoma , including detection of immunogenicity.
* To evaluate pharmacokinetics and pharmacodynamics profiles of AVE1642 as single agent or any PK interactions when given in combination with other anti-cancer therapies.
* To assess the preliminary clinical activity in terms of response rate (Complete response + Partial response), duration of responses, stabilisation rate and duration of stabilisation, according to RECIST criteria.
* To assess the biological activity at the tumor level.

DETAILED DESCRIPTION:
AVE1642 will be administered as an IV infusion on day 1 and then every 3 weeks for at least 2 infusions for evaluability requirements. Curative and / or prophylactic management of allergic reactions during infusion will be implemented when needed. The duration of the study for one patient will include a period for inclusion of up to 2 weeks, at least 2 cycles of treatment in dose escalation step (one cycle of AVE1642 alone and at least one cycle of AVE1642 in combination) and at least one cycle of the combination in the extension cohort, followed, when possible, by a minimum of 30-day follow-up after the last drug administration, in order to detect any potential immunogenicity. In the second step, the patients will continue treatment until disease progression, unacceptable toxicity or willingness to stop.

The expected enrolment period is 15 months with at least 30 day follow-up after the last patient treated.

ELIGIBILITY:
Inclusion Criteria:

* Patients not eligible for surgical resection, liver transplantation, local ablation techniques or chemoembolisation and with histologically proven liver carcinoma whenever possible or combination of radiologically documented hypervascular liver tumour and α foeto protein level ≥ 400 ng/ml
* Signed and dated approved patient informed consent form prior to enrollment into the study

Exclusion Criteria:

* ECOG performance status > 2
* Inadequate organ function:

  * Neutrophils (ANC) < 1,500/mm3
  * Hemoglobin < 10g/dl
  * Platelets < 100,000/mm3
  * Total bilirubin > 1.5 x ULN
  * ASAT, ALAT > 3 x ULN
  * Creatininemia > 1.5 x ULN (or ≥ 2.0 mg/dl)
  * INR > 1.6
  * Liver cirrhosis Child Pugh B or C (score > 6)
  * HbA1C > 8%
* No measurable or evaluable tumoral lesion
* Patients not eligible for sorafenib therapy and for whom this therapy cannot be postponed by 3 weeks (during AVE1642 single treatment period) in dose escalation part
* Prior exposure to an anti-IGF-1R class compound

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) based on grade = or > 3 hematological or non-hematological toxicity and on fasting hyperglycemia | Cycle 1 and cycle 2 (6 weeks)

SECONDARY OUTCOMES:
Anti tumoral activity | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rosmorduc, Professor, Principal Investigator — Hôpital St Antoine, 184 rue du Faubourg St Antoine, 75012 Paris - France
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France